CLINICAL TRIAL: NCT05526274
Title: Clinical Epidemiology of Non-alcoholic Fatty Liver Disease in Children and Adolescents. The LiverKids Study.
Brief Title: Clinical Epidemiology of NAFLD in Children and Adolescents
Acronym: LiverKids
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Hospital del Mar Research Institute (IMIM) (Other); Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other); Fundació Institut Germans Trias i Pujol (Other)
Responsible Party: Sponsor
Other Study IDs: SLT/21/000047
Record Dates: First submitted 2022-08-29; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Childhood Obesity
Keywords: Vibration-Controlled Transient Elastography; Controlled Attenuation Parameter; Lifestyle; Liver fibrosis; Primary care
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Pediatric Obesity; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Analytical determination will be performed on all subjects, after 12 hours of fasting, at the Primary Care Centre. It will include:
  1. blood count, glucose, glycosylated haemoglobin, basal insulin levels, total cholesterol, high-density lipoprotein(HDL-cholesterol), low-density lipoprotein(LDL-cholesterol), triglycerides(TG), transaminases (AST, ALT), gamma-glutamyl-transpeptidase(GGT), alkaline phosphatase, total bilirubin, sideremia, transferrin, transferrin saturation index, total protein, albumin, urea, creatinine, sodium, potassium, TSH and T4.
  2. Determination of insulin resistance using the HOMA method: blood glucose(mmol/L) x insulin(mU/L)/22,5.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General population aged ≥9 to ≤16 years.
  Interventions: Diagnostic Test: Vibration-Controlled Transient Elastography (VCTE) with Controlled Attenuation Parameter (CAP)

INTERVENTIONS:
Diagnostic Test: Vibration-Controlled Transient Elastography (VCTE) with Controlled Attenuation Parameter (CAP) — VCTE with associated CAP is an effective, non-invasive and safe diagnostic method to estimate the degree of fibrosis and steatosis in the liver.

SUMMARY:
Background: Non-alcoholic fatty liver disease (NAFLD) is rapidly increasing alongside overweight and obesity, not only in adults but also in children and adolescents. It is unknown what impact the development of NAFLD in childhood may have in later life. The importance of early detection and treatment lies in its potential for progression to cirrhosis, liver cancer and liver-related death, as well as its associated extrahepatic comorbidities. Vibration-Controlled Transient Elastography (VCTE) with Controlled Attenuation Parameter (CAP) is an effective, non-invasive and safe diagnostic method to estimate the degree of fibrosis and steatosis in the liver, but little is known about its applicability in the paediatric population. Objectives: 1) To assess the prevalence of significant liver fibrosis (LSM≥6,5kPa) using VCTE, and that of non-alcoholic fatty liver disease (≥225dB/m) using CAP in children and adolescents. 2) To determine the optimal cut-off points of the CAP to achieve maximum concordance with the Magnetic Resonance Imaging (MRI) findings in the diagnosis of mild, moderate and severe NAFLD in children and adolescents. Methods: cross-sectional population-based study which will include 2.866 subjects aged ≥9 to ≤16 years. Participants will undergo: anamnesis, physical examination, blood extraction, VCTE, MRI and questionnaires on socio-demographic data, personal and family medical history and lifestyle assessment. Applicability and relevance: the study aims to establish the foundations for the use of VCTE in children and adolescents in order to achieve early diagnosis of NAFLD. Moreover, it will serve to understand in further detail the disease and to identify the risk groups of children and adolescents who may be at risk of developing it. Ultimately, this will help determine to which subgroups of the population we need to target resources for prevention and early detection of this entity, as well as possible intervention for its treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 9 and 16 years.
* Subjects whose parents/legal guardians have signed the informed consent.
* For subjects over 12 years: it will also be necessary to have their own signed informed consent.

Exclusion Criteria:

* Subjects with previously diagnosed liver disease.
* Subjects receiving hepatotoxic drug treatment.
* Subjects with diagnosed eating disorders.

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will be carried out among children and adolescents aged between 9 and 16 years who are enrolled in the Spanish compulsory education system in the territory of Mataró. Since schooling at state level is compulsory in this age group, more than 90% of this population will be accessible from the schools themselves.
Sampling Method: Probability Sample
Enrollment: 2866 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with LSM ≥6.5 kPa by VCTE in the general population aged ≥9 to ≤16 years | 2022-2024
Percentage of subjects with CAP ≥225 dB/m by VCTE in the general population aged ≥9 to ≤16 years. | 2022-2024
Comparison of liver steatosis diagnosis accuracy between CAP by VCTE and MRI in the general population aged ≥9 to ≤16 years. | 2022-2024
Determination of optimal cut-off points of the CAP for the diagnosis of mild, moderate and severe liver steatosis in children and adolescents. | 2022-2024

SECONDARY OUTCOMES:
Comparison of liver steatosis diagnosis accuracy between CAP by VCTE and Fatty Liver Index (FLI) in the general population aged ≥9 to ≤16 years | 2022-2024
Comparison of liver fibrosis diagnosis accuracy between LSM by VCTE and two fibrosis scores (Pediatric NAFLD Fibrosis Index and Pediatric NAFLD Fibrosis Score) in the general population aged ≥9 to ≤16 years | 2022-2024
Detection and structuring of the variables that constitute a specific biomarker for the paediatric-juvenile population that is capable of accurately determining the presence of hepatic steatosis | 2022-2024
Correlation of liver steatosis diagnosis using CAP by VCTE or FLI with the presence of lifestyle and socio-economic factors associated with NAFLD in the general population aged ≥9 to ≤16 years | 2022-2024
Percentage of subjects with BMI ≥30 in the general population aged ≥9 to ≤16 years | 2022-2024
Percentage of subjects with Metabolic Syndrome according to the International Diabetes Federation (IDF) consensus criteria for children and adolescents in the general population aged ≥9 to ≤16 years. | 2022-2024

CONTACTS AND LOCATIONS:
Locations (1):
- IDIAP Jordi Gol i Gurina, Mataró, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chacon C, Arteaga I, Martinez-Escude A, Ruiz Rojano I, Lamonja-Vicente N, Caballeria L, Ribatallada Diez AM, Schroder H, Montraveta M, Bovo MV, Gines P, Pera G, Diez-Fadrique G, Pachon-Camacho A, Alonso N, Graupera I, Toran-Monserrat P, Exposito C. Clinical epidemiology of non-alcoholic fatty liver disease in children and adolescents. The LiverKids: Study protocol. PLoS One. 2023 Oct 13;18(10):e0286586. doi: 10.1371/journal.pone.0286586. eCollection 2023. PMID 37831682